CLINICAL TRIAL: NCT05743010
Title: A Phase 1b Randomized, Double-blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of APL-1401 in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Phase 1b Study to Evaluate APL-1401 in Patients With Moderately to Severely Active Ulcerative Colitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Yahong Meditech Co., Ltd aka Asieris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YHGT-UC-01
Record Dates: First submitted 2022-11-15; First posted 2023-02-24 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — nepicastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APL-1401 (Experimental): On Day 1, patients will be randomized to receive either APL-1401 or placebo in a 5:1 ratio. Patients will receive APL-1401 orally once daily (QD) during the 28-day treatment period.
  Interventions: Drug: APL-1401
- Placebo (Placebo Comparator): Identically matching placebo capsules once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: APL-1401 — APL-1401 capsules orally once daily
  Other Names: Nepicastat; SYN117
  Arms: APL-1401
Drug: Placebo — Placebo capsules orally once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase 1b study designed to evaluate safety, tolerability, PK, and preliminary efficacy of APL-1401 in patients with moderately to severely active UC. This study comprises 3 periods including screening period (D-28~D-1), treatment period (D1-D28), and safety follow-up period(D29-D58).

DETAILED DESCRIPTION:
On Day 1, patients who meet all entry criteria and none of the exclusion criteria will be randomized to receive either APL-1401 or placebo in a 5:1 ratio. Patients will receive APL-1401 orally once daily (QD) during the 28-day treatment period.

Three cohorts with increasing doses of APL-1401 will be explored. The dose of APL-1401 will start at 120 mg QD in Cohort 1 and sequentially increase to 160 mg QD and 200 mg QD in Cohort 2 and Cohort 3, respectively. Three cohorts with increasing doses of APL-1401 will be explored. 200mg QD is designed to be maximum dose in this study.

In one cohort, if dose stopping criteria of cohort is not met, Safety Monitoring Committee (SMC) will be held when last patient completes 28-day of study treatment. SMC will determine whether to continue the study to next cohort base on pre-defined dose escalation criteria, safety data, and available PK data. At this dose strength, if patients are well tolerated and SMC decides to escalate to a higher dose, the next cohort will be started.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Age 18-65 years (inclusive).
3. With a history of UC diagnosis at least 3 months prior to screening.
4. Currently has active UC, defined as a Total Mayo Score of 6 to 12 (inclusive), at baseline, and with a Mayo Endoscopic Sub-Score (MESS) ≥ 2 confirmed by a site reader.
5. Has a rectal bleeding score ≥1 and a stool frequency Score ≥1 and in addition to MESS ≥2 during screening.
6. May be receiving the following drugs:

   1. Oral 5-ammosahcylate (5-ASA) class of medications (mesalamine, olsalazine, balsalazide, sulfasalazine), provided the prescribed dose has been stable for at least 4 weeks prior to randomization; dose must be stable during the treatment period.
   2. Oral corticosteroid therapy (prednisone prescribed at a stable dose ≤ 30 mg/day or budesonide prescribed at a stable dose of ≤ 9 mg/day), provided the prescribed dose has been stable for at least 2 weeks prior to randomization; during the treatment period, the same dose should be maintained but can be tapered by the investigators.
7. Women of childbearing potential must have a negative pregnancy test at screening visit and agree to use 2 highly effective methods of birth control at the same time during entire study period.
8. Male subjects must agree to use protocol specified method(s) of contraception from screening visit until 3 months after last dose.

Exclusion Criteria:

1. Has fulminant colitis, toxic megacolon, primary sclerosing cholangitis, Crohn's disease, history of colitis-associated colonic dysplasia, active peptic ulcer disease.
2. Has a current clinically significant bacterial, parasitic, fungal, or viral infection.
3. Is positive for hepatitis A, B or C, human immunodeficiency virus (HIV), or tuberculosis.
4. Uses any of the following medications:

   1. Intravenous corticosteroids 1 week prior to randomization;
   2. Topical 5-ASA compounds or topical steroid (i.e., enemas or suppositories) 2 weeks prior to randomization;
   3. Anti-diarrheal medications 2 weeks prior to randomization;
   4. Sphingosine 1-phosphate receptor (S1PR) modulator including ozanimod 9 prior to randomization;
   5. JAK inhibitors including tofacitinib and upadacitinib 4 weeks prior to randomization;
   6. TNF-α antagonist including (but not limited to) infliximab, adalimumab, golimumab, certolizumab, or biosimilar agents 10 weeks prior to randomization;
   7. Integrin antagonist, including vedolizumab 18 weeks prior to screening and natalizumab 10 weeks prior to screening;
   8. Interleukin antagonist including ustekinumab 14 weeks prior to screening;
   9. Patients receiving any of the following medications, if they were not discontinued at least 2 weeks prior to randomization: azathioprine, 6-mercaptopurine, methotrexate, mycophenolate mofetil, cyclosporine, tacrolimus, sirolimus, thalidomide. See Table 1;
   10. Prohibited concomitant medications as described in Section 6.5.2 Table 1.
5. Participated in another clinical study of an investigational drug (or medical device) within 30 days prior to screening or is currently participating in another study of an investigational drug (or medical device).
6. Has clinically significant abnormalities in laboratory tests (complete blood count, chemistry panel, TSH, total T3, free T4, urinalysis

   1. Hepatic panel (AST, ALT, total bilirubin) >2 times the upper limits of normal (ULN)
   2. Estimated CrCl <60 mL/min as calculated by the Cockcroft-Gault equation
   3. Thyroid stimulating hormone (TSH) <2.5 mIU/L or >4.2 mIU/L
7. Has a resting heart rate (HR) of <50 bpm or >120 bpm.
8. Has a resting systolic blood pressure >160 mmHg or <90 mmHg.
9. With thyroid disease or history thyroid surgery or on thyroid medications
10. Has orthostatic hypotension (decrease in systolic blood pressure >20 mmHg or decrease in diastolic blood pressure >10 mmHg when going from supine to standing) or a history of clinically significant orthostatic dizziness.
11. Treatment with Class Ia or Class III anti-arrhythmic drugs or treatment with two or more agents in combination known to prolong PR interval.
12. Is taking concomitant beta-blockers (including ophthalmologic timolol), amiodarone, reserpine, clonidine, monoamine oxidase (MAO) inhibitors, alpha blocking drugs, vasodilators which could enhance the production of catecholamines (hydralazine and nitrates), substrates or inhibitors of N-acetyltransferase.
13. Alcohol abuse or alcohol dependence at least 3 months prior to first dose.
14. With history of drug-related rash or has clinically significant rash or pruritus.
15. Has severe COVID-19 infection and needs to use ventilator or other treatments that make using of study drug impossible.
16. With moderate to severe (Child-Pugh Class B and Class C) hepatic impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants adverse events (AEs) | Up to 30 days after the last dose
  An AE was defined as any untoward and unintended medical experience (sign, symptom, appearance of new illness or deterioration of pre-existed disease, abnormal laboratory finding or other medical event) in a patient from obtaining informed consent form, but which did not necessarily have a causal relationship with the study intervention.
  Incidence of serious adverse events (SAEs) Incidence of adverse events leading to investigational drug discontinuation Incidence of adverse events of special interest (AESI) Laboratory evaluation results Vital sign measurements Physical examination findings
Number of Participants serious adverse events (SAEs) | Up to 30 days after the last dose
  An SAE is defined as any untoward medical occurrence that, at any dose, including results in death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, a congenital anomaly/birth defect, other situations.
Number of Participants adverse events of special interest (AESI) | Up to 30 days after the last dose
  An adverse event of special interest (AESI) is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor is required, including rash, orthostatic hypotension, thyroid dysfunction.

SECONDARY OUTCOMES:
Cmax | Day 1 through Day 28
  Maximum observed plasma concentration
Tmax | Day 1 through Day 28
  Time to maximum plasma concentration
T1/2 | Day 1 through Day 28
  Plasma half-life
AUClast | Day 1 through Day 28
  Area under the plasma concentration-time curve from 0 to last measurable concentration
AUC0-24 | Day 1 through Day 28
  Area under the plasma concentration-time curve from 0 to 24 hours
AUC | Day 1 through Day 28
  Area under the plasma concentration-time curve from 0 to infinity
Cave | Day 1 through Day 28
  Average plasma concentration (steady state)
Cmin | Day 1 through Day 28
  Minimum plasma concentration at time of dosing (steady state)
Cmax/Cmin | Day 1 through Day 28
  Peak to minimum plasma concentration (steady state)
Cmax/Cave | Day 1 through Day 28
  Peak to average plasma concentration (steady state)
Fluctuation | Day 1 through Day 28
  100 (Cmax-Cmin)/Cave-percent fluctuation about average plasma concentration (steady state)
Clinical response | Day 1 through Day 28
  Clinical response, as assessed by Mayo Score, defined as a decrease from baseline in Total Mayo Score of ≥3 points and ≥30%, and a decrease from baseline in the rectal bleeding sub-score of ≥1 point or an absolute rectal bleeding sub-score of 0 or 1 point, after 28 days of treatment compared to baseline.
  The Mayo Score is a composite index of four items (stool frequency, rectal bleeding, endoscopy findings, and physician's global assessment) with each item graded semi-quantitatively on a scale of 0 to 3 where 0 represents normal and higher score represents more severe disease status. The total Mayo Score is the sum of the four item scores, with a result ranging from 0 to 12 points. Higher scores represent more severe disease.
Endoscopic improvement | Day 1 through Day 28
  Endoscopic improvement, as assessed by the endoscopic sub-score of the Total Mayo Score, defined as an endoscopy sub-score of 0 or 1 point, after 28 days of treatment compared to baseline.
Histologic remission | Day 1 through Day 28
  Histologic remission, as assessed by Geboes Score, defined as a Geboes Score <2.0, after 28 days of treatment compared to baseline.

OTHER OUTCOMES:
CRP | Day 1 through Day 28
  Plasma biomarker: plasma C reactive protein (CRP)
ESR | Day 1 through Day 28
  Plasma biomarker: plasma erythrocyte sedimentation rate (ESR)
Fecal lactoferrin | Day 1 through Day 28
  Stool biomarker: faecal lactoferrin
Fecal calprotectin | Day 1 through Day 28
  Stool biomarker: fecal calprotectin

CONTACTS AND LOCATIONS:
Overall Officials: Qiuyue QU, Study Director — Jiangsu Yahong Meditech Co., Ltd aka Asieris
Locations (4):
- United States (4):
  - New Hope Research Development, Corona, California
  - Guardian Angel Research Center, Tampa, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Meridian Clinical Research, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No